CLINICAL TRIAL: NCT04105140
Title: Oxytocin Effects on the Prosocial Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-44
Record Dates: First submitted 2018-09-09; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: oxytocin; prosocial learning
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- male oxytocin group (Experimental): male subjects with oxytocin treatment
  Interventions: Drug: Oxytocin
- male placebo group (Placebo Comparator): male subjects with placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — intranasal administration of oxytocin (24 IU)
  Arms: male oxytocin group
Drug: Placebo — intranasal administration of placebo (24 IU)
  Arms: male placebo group

SUMMARY:
To investigate whether intranasal oxytocin (24 IU) treatment can influence prosocial learning behavior in males.

DETAILED DESCRIPTION:
In a double-blind, within-subject, placebo controlled design, investigators plan to investigate the effect of oxytocin treatment on prosocial learning. Before the self-administration, participants need to finish several questionnaires including IRI, AAS, BASBIS, SPSRQ, SES, PTM, STAI, BDI, ASQ and PNAS. They would finish the PANAS again before the scanning.

Participants are informed that they perform the reward learning task either for themselves, another (unknown) person or no one (control). In the probabilistc reward learning task, associations with two stimuli with different reward probabilities are learned via monetary feedback (reward ￥1 or no reward ￥0). After the experiment, participants need to finish the PANAS.

ELIGIBILITY:
Inclusion Criteria:

* without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Neural processing during feedback based on prosocial learning assessed by fMRI scanner | 1 hour
  fMRI BOLD indices of neural processing learning related brain regions will be compared between the treatment administrations.

SECONDARY OUTCOMES:
Behavioral learning performance measured by E-prime | 1 hour
  Learning performance will be compared between the treatment administrations by calculating the accuracy of learning.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China